CLINICAL TRIAL: NCT05384288
Title: Response to Influenza Vaccination in Pediatric Oncology Patients
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RIVIPOP; NCI-2022-05167 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancy; Pediatric Cancer; Transplant-Related Cancer
Keywords: Influenza infection
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Pediatric Influenza Vaccine Recipients: Pediatric patients eligible to receive seasonal influenza vaccine.

SUMMARY:
Influenza infection occurring during oncologic treatment or following hematopoietic cell transplantation (HCT) is associated with increased risk of morbidity in the form of lower respiratory tract infection (LRTI) and mortality relative to otherwise healthy patients. The study participants have been diagnosed with a hematological malignancy and are eligible to receive the current seasonal influenza (Flu) vaccine.

Primary Objective

* To determine the feasibility of opening a longitudinal prospective study of IIV immunogenicity in pediatric leukemia patients.
* To describe the immunogenicity, as measured by the development of cell- and/or antibody-mediated influenza specific responses 3 to 5 weeks following vaccination, in a cohort of pediatric leukemia patients.

Secondary Objectives

* To describe whether an immune response, as measured by development of cell- and/or antibody-mediated influenza specific responses, is detectable 1-2 weeks following vaccination in a cohort of pediatric leukemia patients.
* To describe the durability of immunogenicity by measuring cell - and antibody- mediated influenza specific responses at 6 months and 1 year following vaccination in a cohort of pediatric leukemia patients.

Exploratory Objectives

* To estimate the clinical effectiveness of influenza vaccine in this cohort by monitoring for the development of clinical diagnosis of influenza in the cohort of enrolled pediatric oncology patients.
* To correlate results of immune cell frequency in blood, as measured by complete blood count with differential, with development of an immune response to IIV.

DETAILED DESCRIPTION:
This is a prospective, 2-stage, non-therapeutic study to characterize the immunogenicity of influenza vaccination among pediatric oncology patients at St. Jude. The first stage of the study will consist of a feasibility phase to assess the feasibility of opening a longitudinal prospective study of IIV immunogenicity in pediatric leukemia patients. The second stage will assess the immunogenicity of IIV among pediatric leukemia patients in a larger samples size. The investigator will collect about one teaspoon of blood from the study participant up to 6 times over a year for a total of 6 teaspoons a year. The investigator will also collect some information about the study participant's underlying condition, flu testing and overall health from the medical record during this time.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≤ 18 years old at the time of consent receiving care at St. Jude Children's Research Hospital
* Diagnosed with a hematological malignancy
* Eligible to receive the current seasonal influenza vaccine

Exclusion Criteria:

• Previously received at least one dose of the current seasonal influenza vaccine.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All participants who meet eligible criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of evaluable participants. | 3 years
  Feasibility is estimated as the proportion of evaluable patients who provide a baseline and Day +35 sample. A 95% confidence interval will be provided.
Proportion of participants with immunogenicity 3 to 5 weeks following vaccination. | 3 years
  Immunogenecity will be measured by the development of cell- and antibody-mediated influenza specific responses 3 to 5 weeks following vaccination. Immunogenicity is estimated as the proportion of evaluable patients whose cell- (as measured by development of any detectable specific T cell responses) and antibody-mediated influenza specific responses (as measured by detectable post vaccination antibody titers) 3 to 5 weeks following vaccination. 95% confidence intervals will be provided.

SECONDARY OUTCOMES:
Proportion of participants with an immune response 1 to 2 weeks following vaccination. | 3 years
  The proportion of patients who have detectable cell- and antibody-mediated influenza specific responses 1-2 weeks following vaccination will be estimated along with a 95% confidence interval.
Proportion of participants with durability of immunogenicity at 6 months and 1 year post-vaccination. | 3 years
  The proportion of patients who still have detectable cell- and antibody-mediated influenza specific responses 6 months and 1 year following vaccination will be estimated, respectively. 95% confidence intervals will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Ramilo Octavio, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols